CLINICAL TRIAL: NCT03051724
Title: Telemedicine for CPAP Therapy Control in OSA Patients With Limited Internet Knowledge
Brief Title: Telemedicine for CPAP Therapy Control in OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Jose M. Montserrat, Medical Doctor, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI14/00416_1
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: OSA
Keywords: OSA; CPAP management; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): These OSA patient's are not familiarized with the use of internet and mobile technologies and with CPAP prescription. They follow the intervetion follow up that consists in an adaptation session where the tecnitian delivers them an automatic CPAP machine. Patient's are titrated with this automatic device in 5-7 days and are treated with the automatic device during 3 months.
  The other part of the follow up consists on a voicemail where the patient can contact us 24h a day and on an , with an internet-connected tablet with a special app where the patient's answer a questionnaire once two weeks.
  Interventions: Other: Telematic follow up
- Control group (No Intervention): These patient's are patient's that follow the process that all patient's take during CPAP treatment. During the three months of study, the follow up will be the usual.

INTERVENTIONS:
Other: Telematic follow up — Follow-up of OSA patients through automatic CPAP with data transmission (Dreamstation; Philips Respironics), a 24-hour voice mailbox available for questions or problems, and an Internet-connected (4G) tablet with a friendly mobile application for simple questionnaires.
  Arms: Intervention group

SUMMARY:
Obstructive sleep apnea is a very frequent syndrome and Continuous Positive Airway Pressure (CPAP) is the gold standard treatment. Nevertheless, obtaining the sufficient compliance is complex. New communication technologies and the current health challenges, such as aging and high health care costs have encouraged the interest in new strategies.

As showed recently, telemedicine is an alternative (Isetta, Thorax 2015) in patients that use internet and mobile technologies usually. However, there is a significant percentage of patients that does not use Internet and mobile technologies, only the 58% of patients over 65 years uses them (Dorsey, NEJM 2016). Although evidence regarding telemedicine is conflicting, it suggest that it's applicability depends in patient's characteristics and it is necessary to personalize it to make it safe and effective (Takahashi, Arch Intern Med 2012). That's why the investigators believe that the next step should be to choose those patient's that doesn't use Internet or mobile technologies and to verify the applicability of a telematic system that could facilitate the extra hospital management of this patient's.

The aim of the study is to evaluate the telematic management of various outcomes that are emitted by CPAP machine, and by an app where the patient's will answer different questions regarding their treatment during the three months of study period.

DETAILED DESCRIPTION:
We include OSA patient's that are not familiarized with the use of internet and mobile technologies and with CPAP prescription. They follow up an adaptation session where an automatic CPAP machine is delivered. Patient's are titrated with this automatic device in 5-7 days and are treated with the automatic device during 3 months.

The other part of the follow up consists on a voicemail where the patient can contact the sleep unit 24h a day and on a tablet, with an special app where the patient's answer a questionnaire once two weeks.

ELIGIBILITY:
Inclusion Criteria:

* OSA diagnosis and CPAP prescription
* No use of internet or mobile devices

Exclusion Criteria:

* Unstable diseases and severe comorbidities
* Previous CPAP treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the telematic CPAP follow up | 3 months
  CPAP adherence: Hours of use

SECONDARY OUTCOMES:
Efficacy of titration and follow up of data transmitted by CPAP | 3 months
  Leaks, Residual events
Evaluate the effects of treatment in patient's symptomatology | 3 months
  Epworth questionnaire
Evaluate the satisfaction of patient's and professionals | 3 months
  Satisfaction questionnaire
Evaluate the effect of CPAP treatment and telematic follow up | 3 months
  EQ5D questionnaire
To compare the cost of the telematic follow up group vs hospital group | 3 months
  Bayesian cost analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No